CLINICAL TRIAL: NCT01374399
Title: Effects of an One-year Physical Exercise Intervention on Prognosis, Side-effects and Complications After Allogeneic Stem Cell Transplantation
Brief Title: Physical Exercise Therapy vs Relaxation in Allogeneic Stem Cell Transplantation (PETRA)
Acronym: PETRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other); University Hospital Heidelberg (Other); Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DJCLS R 10/42pf
Record Dates: First submitted 2011-04-18; First posted 2011-06-16 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: allogeneic stem cell transplantation; exercise; survival; fatigue; quality of life; cancer; physical performance
MeSH Terms: conditions — Motor Activity; Fatigue; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- resistance and endurance exercise (Experimental)
  Interventions: Behavioral: exercise and relaxation
- relaxation (Active Comparator)
  Interventions: Behavioral: exercise and relaxation

INTERVENTIONS:
Behavioral: exercise and relaxation — resistance and endurance exercise, 3-5 times per week

SUMMARY:
The PETRA-Study is a randomized, controlled trial and designed to examine the effects of an one-year physical exercise intervention on prognosis, side-effects and complications after allogeneic stem cell transplantation.

The exercise intervention includes both, resistance and endurance training. Patients assigned to the control group perform a relaxation program (progressive muscle relaxation - Jacobsen) and have the same frequency of social contact.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication: allogeneic stem cell transplantation

Exclusion Criteria:

* Orthopeadic limitations that hamper the exercise intervention
* Osseous degenerations that have an improved fracture risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | two years

SECONDARY OUTCOMES:
Fatigue | admission to hospital for allo-HSCT, discharge from hospital (expected average of 4 to 5 weeks after admission), day 100, day 180, day 270 and day 365 post transplanation
  measured by the Multidimensional Fatique Inventory (MFI)
Quality of Life | admission to hospital for allo-HSCT, discharge from hospital (expected average of 4 to 5 weeks after admission), day 100, day 180, day 270 and day 365 post transplanation
  mesured by the European Organistion for Research and Treatment of Cancer questionnaire including the high dose chemotherapy module (EORTC-QLQ-C30/HDC-29)
Hemoglobin, Leukocytes, Thrombocytes | during hospitalisation for allo-HSCT (expected average 4-5 weeks), day 100, day 180, day 270, day 365 post transplantation
  Hematological and immunological reconstitution
Side-effects (Infections, GvHD, Depression, Distress) | during hospitalisation for allo-HSCT (expected average 4-5 weeks), day 100, day 180, day 270, day 365 post transplantation
  Depression mesured by "Allgemeine Depressionskala" (ADS, the German version of the Center for Epidemiological Studies Depression Scale (CES-D)) Distress mesures by the NCCN Distress Thermometer
Adherence to exercise protocol | one year
  Fesability of an one-year exercise intervention after allogeneic HSCT
Muscular strength | admission to hospital for allo-HSCT, discharge from hospital (expected average of 4 to 5 weeks after admission), day 100, day 180, day 270 and day 365 post transplanation
  measured at the IsoMed2000 and/or Handheld Dynamometer
cardiorespiratory fitness | admission to hospital for allo-HSCT, discharge from hospital (expected average of 4 to 5 weeks after admission), day 100, day 180, day 270 and day 365 post transplanation
  measured by ergospirometry (VO2max) and/or 6 Minutes Walk Test (meters)
IL-6, IL-4, IL-8, IL-10, IL-1ra, TNF-alpha, Prostaglandin | admission to hospital for allo-HSCT, discharge from hospital (expected average of 4 to 5 weeks after admission), day 100, day 180, day 270 and day 365 post transplanation
  Biomarker in blood and urine
median survival, non-relapse mortality | admission to hospital until 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bohus, Prof. MD, Principal Investigator — Central Institute of Mental Health; Joachim Wiskemann, PhD, Principal Investigator — National Center for Tumor Diseases; Dreger Peter, Prof. MD, Study Chair — University Hospital Heidelberg
Locations (1):
- German Cancer Research Center, Heidleberg, Germany

REFERENCES:
- [Derived] Limbach M, Kuehl R, Koeppel M, Dreger P, Luft T, Bohus M, Wiskemann J. Factors affecting pretransplant muscle strength in allogeneic stem cell transplant candidates prior transplantation. Support Care Cancer. 2025 Jan 10;33(2):89. doi: 10.1007/s00520-024-09140-8. PMID 39794666
- [Derived] Aziz JA, Smith C, Slobodian M, Du I, Shorr R, De Lisio M, Allan DS. Impact of Exercise Training on Hematological Outcomes Following Hematopoietic Cell Transplantation: A Scoping Review. Clin Invest Med. 2021 Jun 14;44(2):E19-26. doi: 10.25011/cim.v44i2.36369. PMID 34152703
- [Derived] Wiskemann J, Kuehl R, Dreger P, Huber G, Kleindienst N, Ulrich CM, Bohus M. Physical Exercise Training versus Relaxation in Allogeneic stem cell transplantation (PETRA Study) - Rationale and design of a randomized trial to evaluate a yearlong exercise intervention on overall survival and side-effects after allogeneic stem cell transplantation. BMC Cancer. 2015 Sep 7;15:619. doi: 10.1186/s12885-015-1631-0. PMID 26345187